CLINICAL TRIAL: NCT01547637
Title: Preventing the Obturator Nerve Reflex: A Comparison of Ultrasound Guided Obturator Nerve Block and Classic Anatomic Block Technique.
Brief Title: Preventing the Obturator Nerve Reflex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jonathan Anson, Assitant professor of Anesthesiology, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRAMS039186EP
Record Dates: First submitted 2012-02-29; First posted 2012-03-08 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Bladder Injury
Keywords: Obturator nerve block; Regional anesthesia; TURBT

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound Guided (Experimental): Ultrasound guided obturator nerve block will be performed after induction of general anesthesia. The anterior and posterior divisions of the obturator nerve will be identified with ultrasound. A stimulating needle will be inserted under direct ultrasound visualization. The anterior division will be blocked first. When adductor twitches are present at less than or equal to 0.5 mA, 10 ml of 2% lidocaine will be injected. Next, the needle will be re-directed under direct ultrasound visualization towards the posterior branch of the obturator nerve. After twitches < 0.5 mA are achieved then 10 mL of 2% lidocaine will be injected when the needle tip is visualized in proximity of the posterior branch.
  Interventions: Procedure: Obturator nerve block
- Anatomic landmark (Experimental): Obturator nerve block will be performed after induction of general anesthesia. The adductor magnus tendon approach will be used. A 4 cm insulated stimulating needle will be used to verify location of the obturator nerve by contraction of the thigh adductor group. The needle will be advanced until nerve stimulation is still present at less than or equal to 0.5 mA. When the appropriate nerve stimulation is achieved 10 ml of 2% lidocaine will be injected in divided doses with frequent aspiration. Nerve conduction studies will be repeated once a minute for the first 10 minutes after block completion.
  Interventions: Procedure: Obturator nerve block

INTERVENTIONS:
Procedure: Obturator nerve block — Peripheral obturator nerve block using 10 ml of 2% lidocaine
  Other Names: anatomic obturator block
  Arms: Anatomic landmark
Procedure: Obturator nerve block — Ultrasound guided peripheral obturator nerve block
  Other Names: ultrasound guided obturator nerve block
  Arms: Ultrasound Guided

SUMMARY:
The key objective of this study is to compare success rates of ultrasound guided obturator nerve block and anatomic landmark guided obturator nerve block as determined by neuromonitoring endpoints and surgeon observations.

DETAILED DESCRIPTION:
Transurethral resection of bladder tumor (TURBT) is a urologic surgery used in the treatment of non-muscle invasive bladder cancer. A potential complication of this procedure is bladder rupture or injury secondary to adductor muscle contraction from obturator nerve stimulation. This risk is increased in resection of lateral wall tumors, as electrosurgical resection of these lesions is more likely to inadvertently stimulate the obturator nerve.

There are several mechanisms for preventing the obturator reflex. Pharmacologic paralysis can reliably inhibit thigh adduction. However, TURBT is often a short procedure that is not amendable to intermediate duration neuromuscular blocking medications. The use of succinylcholine is another option but is limited by its short duration of action which may not be adequate for the time needed to resect the tumor. Additionally, many patients have contraindications to the use of succinylcholine. Spinal anesthesia does not reliably prevent the obturator reflex.

Regional anesthesia is another potential treatment modality to prevent the obturator reflex during TURBT. Motor blockade of the obturator nerve will prevent this adduction in the event of inadvertent nerve stimulation. Peripheral blockade of the obturator nerve can be combined with either general or spinal anesthesia. Historically, obturator nerve block (ONB) has been considered a technically challenging procedure. Recently, however, successful ultrasound guided ONB techniques have been reported. To the best of our knowledge there has been no study to date comparing the effectiveness of ONB achieved by anatomic landmarks (with nerve stimulation) versus ultrasound guided ONB (with nerve stimulation) at preventing the obturator reflex during TURBT surgery.

The key objective of this study is to compare success rates of ultrasound guided obturator nerve block and anatomic guided obturator nerve block as determined by neuromonitoring endpoints and surgeon observations.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing TURBT for lateral wall bladder tumors at risk for electrical stimulation as determined by the attending surgeon.

Exclusion Criteria:

* Pre-existing obturator nerve injury
* Thigh adductor muscle weakness
* Neuropathy
* Local anesthetic allergy
* Infection at the site of injection
* Abnormal coagulation studies
* use of neuromuscular blocking medications (if deemed necessary by attending anesthesiologist caring for the patient).

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-05; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Nerve conduction velocity | 1 day
  Neuromonitoring technician will measure and record obturator nerve conduction velocity in pre-defined time intervals after performance of obturator nerve block.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan A Anson, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States